CLINICAL TRIAL: NCT07086716
Title: The Role of Frailty in the Rehabilitation Pathway Following Hip or Knee Arthroplasty Surgery.
Brief Title: Frailty in Hip or Knee Arthroplasty Patients.
Acronym: FRAKH
Status: Recruiting | Type: Observational
Sponsor: Joel Pollet (Other)
Responsible Party: Sponsor-Investigator, Joel Pollet, Principal Investigator, Fondazione Don Carlo Gnocchi Onlus
Organization: Fondazione Don Carlo Gnocchi Onlus (Other)
Other Study IDs: JP-004
Record Dates: First submitted 2025-07-08; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Frail Elderly; Arthroplasties Hip Replacement; Arthroplasty Knee
Keywords: Frailty; Hip; Knee; Arthroplasty; rehabilitation
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Frail and Knee Arhtroplasty: Subjects with frailty before receiving knee arthroplasty
- Non-Frail and Knee Arhtroplasty: Subjects without frailty before receiving knee arthroplasty
- Frail and Hip Arhtroplasty: Subjects with frailty before receiving hip arthroplasty
- Non-Frail and Hip Arhtroplasty: Subjects without frailty before receiving hip arthroplasty

SUMMARY:
The study aims to understand the existing differences between frail and non-frail subjects who underwent a rehabilitation path after receiving hip or knee arthroplasty surgery.

DETAILED DESCRIPTION:
This study wanted to investigate the role of frailty in the rehabilitation path following hip or knee arthroplasty. Subjects will be divided according to the type of arthroplasty received (i.e., hip or knee arthroplasty). Consequently, each arthroplasty group will be divided into a frail group and a non-frail group based on the presence of frailty conditions before receiving surgery. Frailty condition will be assessed using the Primary Care Frailty Index, based on the information reported in each patient's medical record before surgery. Frailty level will be reassessed during the rehabilitation period, specifically at hospitalization in the rehabilitation ward (T0) and Discharge (T1). While other time points considered for the primary outcomes will be at 3-month follow-up (T2) and 1-year follow-up (T3), alongside the primary and secondary outcomes chosen for the study. The different outcomes considered in this study were selected to provide a wide range of information regarding body structure and function, activity level, and perceived level of satisfaction with the intervention. Moreover, the long-term follow-up will collect data on the adverse event rate, which previous studies have shown to significantly impact more frail subjects after receiving arthroplasty. However, the possible protective role of rehabilitation has never been considered. This prospective case-control study is the first to consider the crucial role of rehabilitation in the post-surgical path of subjects receiving arthroplasties. It can serve as a preliminary basis for further trials based on tailored interventions for frail subjects.

ELIGIBILITY:
Inclusion Criteria:

* Received elective hip or knee arthroplasty;
* Ability to understand written and oral instructions;
* Gave consent to study participation.

Exclusion Criteria:

* Arthroplasty revision or not elective intervention;
* Participation in other studies;
* Hospitalized in the rehabilitation ward more then 10 days after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will include subjects that after an elective intervention of knee or hip arthroplasty are hospitalized in the thertiary refferal rehabilitation center where we are conducting the study.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Oxford Hip Score | Hospitalization or Day 1 (T0), to the discharge avarege Day 20 (T1), till 3 months after surgery (T2), and 1 year after surgery(T3).
  It'a Patient Reported Outcome specific for patients that received Hip Arthroplasty. It investigates the field of autonomy, participation, and pain.
Oxford Knee Score | Hospitalization or Day 1 (T0), to the discharge avarege Day 20 (T1), till 3 months after surgery (T2), and 1 year after surgery(T3).
  It'a Patient Reported Outcome specific for patients that received Knee Arthroplasty. It investigates the field of autonomy, participation, and pain.

SECONDARY OUTCOMES:
modified Barthel Index | Hospitalization or Day 1 (T0), to the discharge avarege Day 20 (T1).
  Investigates the ability of the included subjects to perform autonomously their Activities of Daily Living
Numerical Pain Raitng Scale | Hospitalization or Day 1 (T0), to the discharge avarege Day 20 (T1), till 3 months after surgery (T2), and 1 year after surgery(T3).
  Provides a value of perceived pain from 0 to 10
Adverse events | Hospitalization or Day 1 (T0), to the discharge avarege Day 20 (T1), till 3 months after surgery (T2), and 1 year after surgery(T3).
  Each adverse events, related to the arthroplasty, occuring to subjects involved in the study will be monitored, in particular: Death, arthroplasty dislocation, joint infection, reoperation, wound healing disorder, periprosthetic fracture, mechanical failure, and heterotopic ossification.
International Knee Society Rating System | Hospitalization or Day 1 (T0), to the discharge avarege Day 20 (T1).
  Rates the functioning of the knee joint, in subjects who underwent Knee arthroplasty
Merlè D'Aubigne-Postel Scale | Hospitalization or Day 1 (T0), to the discharge avarege Day 20 (T1).
  Rates the functioning of the knee joint, in subjects who underwent Hip arthroplasty

OTHER OUTCOMES:
Gait speed | Hospitalization or Day 1 (T0), to the discharge avarege Day 20 (T1).
  Gait speed recorded during gait analysis
Cadence | Hospitalization or Day 1 (T0), to the discharge avarege Day 20 (T1).
  Step cadence recorded during gait analysis
Gait cycle length | Hospitalization or Day 1 (T0), to the discharge avarege Day 20 (T1).
  Step length recorded during gait analysis
Gait cycle duration | Hospitalization or Day 1 (T0), to the discharge avarege Day 20 (T1).
  Step duration recorded during gait analysis
Step subphases duration | Hospitalization or Day 1 (T0), to the discharge avarege Day 20 (T1).
  Duration of single stance, double stance and swing phase recorded through gait analysis.
Gait Profile Score | Hospitalization or Day 1 (T0), to the discharge avarege Day 20 (T1).
  A gait summary measure that indicates the deviation from a physiological gait
Gait Variable Score | Hospitalization or Day 1 (T0), to the discharge avarege Day 20 (T1).
  A gait summary measure that indicates the deviation from physiological motion in the main joint plains of movement.
Gait Deviation Index | Hospitalization or Day 1 (T0), to the discharge avarege Day 20 (T1).
  Provides the deviation rate from physiological gait.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro "E. Spalenza - Don Gnocchi, Rovato, BS, Italy

IPD SHARING:
Plan to Share IPD: Yes
We will upload the anonimazied database of the study in Zenodo (https://zenodo.org/), with a specific indication to the repository in the full-publication.
Supporting Information: Study Protocol
Time Frame: Immediatly following the publication. No end date.
Access Criteria: Anyone who wishes to access the data